CLINICAL TRIAL: NCT00196495
Title: Clinical Assessment of the Total Vaginal Mesh Technique for Treatment of Genital Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003-016
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-12-18 (Estimated); Status verified 2006-12

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

INTERVENTIONS:
Device: Polypropylene Mesh

SUMMARY:
Pelvic floor prolapse is a general term used to describe various clinical conditions that are associated with pelvic floor (muscles that support the vagina) relaxation in female patients.Pelvic floor prolapse is thought to result from a stretching, weakening or tearing of the soft tissue structures that support the pelvic organs. These tissues become compromised because of a weakened or damaged.The purpose of the study will be to demonstrate the usability of Polypropylene Mesh for prolapse repair, using the TVM technique.

ELIGIBILITY:
Inclusion Criteria:

* Female candidate for surgical pelvic floor repair (at least ICS stage II symptomatic prolapse).
* Patient who is at leat 21 years of age.
* Patient whose family is complete.
* Patient may not have uncontrolled diabetes.

Exclusion Criteria:

* Patients may not have coagulation disorders.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-06; Study Completion 2005-11

PRIMARY OUTCOMES:
Effectiveness of the TVM treatment in curing vaginal prolapse as indicated by recurrence rate.

SECONDARY OUTCOMES:
Intraoperative complication
Patient tolerance of the synthetic mesh placed
Postoperative complications
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.